CLINICAL TRIAL: NCT05469984
Title: Comparing Obstetrical Outcomes and Infectious Morbidity Between Two Prophylactic Antibiotic Protocols in Women With Term Prolonged Pre-labor Rupture of Membrane and Preterm Labor
Brief Title: Comparing Two Prophylactic Antibiotic Protocols in Women With Term Prolonged Pre-labor Rupture of Membrane and Preterm Labor
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, Dr. Maya Wolf, Director- Fetal Maternal Medicine Unit, Western Galilee Hospital-Nahariya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0103-22-NHR
Record Dates: First submitted 2022-07-09; First posted 2022-07-22 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Preterm Labor With Preterm Delivery; Premature Rupture of Membranes Prolonged
Keywords: prolonged term PROM; pre-term labor; prophylactic antibiotic; peripartum infection; bacterial distribution
MeSH Terms: interventions — Ampicillin; Gentamicins

STUDY DESIGN:
Intervention Model Description: women with prolonged premature rupture of membrane>18 h or women in preterm delivery will be randomized to receive one of two prophylactic antibiotic treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- women with term prolonged>18h rupture of membrane (Active Comparator): women with term prolonged >18 h prom or in preterm delivery will be treated with IV ampicillin 2 gr every 6 hours until delivery
  Interventions: Drug: Ampicillin Only Product; Drug: ampicillin plus gentamicin
- women with preterm labor (Active Comparator): women with term prolonged >18 h prom or in preterm delivery will be treated with IV ampicillin 2 gr every 6 hours until delivery plus IV gentamicin 5 mg/kg every 24 hours
  Interventions: Drug: Ampicillin Only Product; Drug: ampicillin plus gentamicin

INTERVENTIONS:
Drug: Ampicillin Only Product — women will be randomize to receive Ampicillin Only Product or ampicillin plus gentamicin
Drug: ampicillin plus gentamicin — women will be randomize to receive Ampicillin Only Product or ampicillin plus gentamicin

SUMMARY:
This randomized prospective trial aimed to compare 2 prophylactic antibiotic regiment (ampicillin alone versus ampicillin plus gentamycin) in term prolonged pre-labor rupture of membrane and in preterm deliveries and examine related obstetrical outcome and infectious morbidity

DETAILED DESCRIPTION:
Maternal peripartum fever is a common complication of pregnancy and postpartum period associated with potentially serious obstetrical outcomes and infectious morbidity. Peripartum infections includes intrapartum intraamniotic infection (IAI) and postpartum endometritis. Both are caused by polymicrobial bacterial infection. Increased latency period from rupture of membranes (ROM) until delivery is a common risk factor. Another risk factor is pre-term delivery.

This randomized prospective trial aimed to compare 2 prophylactic antibiotic regiment (ampicillin alone versus ampicillin plus gentamycin) in term prolonged pre-labor rupture of membrane and in preterm deliveries and examine related obstetrical outcome and infectious morbidity.

Primary outcome-peripartum infections- chorioamnionitis, endometritis and surgical site infection secondary outcome- obstetrical outcome- mode of delivery, Apgar score, cord blood pH, peripartum fever, maternal length of admission, postpartum maternal antibiotic treatment, Surface swab cultures were obtained from the placenta, amnion and umbilical cord (birth cultures) and uterine swab cultures, maternal blood culture, placental histologic evaluation neonatal outcomes-NICU admission, length of admission, neonatal morbidity-ventilation support, early neonatal sepsis

ELIGIBILITY:
Inclusion Criteria: maternal age > 18 years singleton pregnancy vertex presentation prolonged >18 h prom or preterm delivery

-

Exclusion Criteria:

* GBS carrier
* preterm premature rupture of membrane for conservative treatment
* intra-uterine fetal death fetal major anomaly
* drug allergy for the antibiotic in use in this study
* women receiving antibiotic treatment for other infection such as urinary tract infection

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — women 18 years or older with singleton pregnancy
Enrollment: 600 (Estimated)
Dates: Start 2022-11-25 (Actual); Primary Completion 2025-09-25 (Estimated); Study Completion 2025-09-26 (Estimated)

PRIMARY OUTCOMES:
endometritis rate | up to 6 weeks postpartum
chorioamnionitis rate | during labor (up to delivery of the newborn)

SECONDARY OUTCOMES:
cord blood pH | immediately after delivery of the placenta
maternal intrapartum fever | during labor (up to delivery of the newborn)
  body temperature,
NICU (neonatal intensive care unit) hospitalization length, | up to 3 month from delivery
  days
rate of neonatal early onset sepsis | up to one week from delivery
  positive blood culture
Rate of participants treated with antibiotics during the postpartum period | 6 week postpartum
maternal postpartum hospitalization length | up to 6 weeks post partum
Number of neonate with ventilation support | one week from delivery
Number of neonate treated with antibiotics | one week from delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Galil Medical Center, Nahariya, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Apantaku O, Mulik V. Maternal intra-partum fever. J Obstet Gynaecol. 2007 Jan;27(1):12-5. doi: 10.1080/01443610601016644. PMID 17365450
- [Background] Committee Opinion No. 712: Intrapartum Management of Intraamniotic Infection. Obstet Gynecol. 2017 Aug;130(2):e95-e101. doi: 10.1097/AOG.0000000000002236. PMID 28742677
- [Background] Kachikis A, Eckert LO, Walker C, Bardaji A, Varricchio F, Lipkind HS, Diouf K, Huang WT, Mataya R, Bittaye M, Cutland C, Boghossian NS, Mallett Moore T, McCall R, King J, Mundle S, Munoz FM, Rouse C, Gravett M, Katikaneni L, Ault K, Klein NP, Roberts DJ, Kochhar S, Chescheir N; Brighton Collaboration Chorioamnionitis Working Group. Chorioamnionitis: Case definition & guidelines for data collection, analysis, and presentation of immunization safety data. Vaccine. 2019 Dec 10;37(52):7610-7622. doi: 10.1016/j.vaccine.2019.05.030. No abstract available. PMID 31783982
- [Background] Yoon BH, Romero R, Moon JB, Shim SS, Kim M, Kim G, Jun JK. Clinical significance of intra-amniotic inflammation in patients with preterm labor and intact membranes. Am J Obstet Gynecol. 2001 Nov;185(5):1130-6. doi: 10.1067/mob.2001.117680. PMID 11717646
- [Background] Soper DE, Mayhall CG, Froggatt JW. Characterization and control of intraamniotic infection in an urban teaching hospital. Am J Obstet Gynecol. 1996 Aug;175(2):304-9; discussion 309-10. doi: 10.1016/s0002-9378(96)70139-4. PMID 8765246